CLINICAL TRIAL: NCT03196557
Title: An Experimental Medicine Study to Assess the Pharmacodynamics Following Administration of Multiple Doses of Prednisolone to Healthy Male Subjects
Brief Title: A Study to Assess the Pharmacodynamics (PD) of Prednisoline in Healthy Male Subject
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IM124-001
Record Dates: First submitted 2017-06-21; First posted 2017-06-22 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Immunoscience

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Specified dose on specified days
  Interventions: Drug: Prenisolone
- Arm B (Placebo Comparator): Specified dose on specified days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prenisolone — Specified dose on specified days
  Arms: Arm A
Drug: Placebo — Specified dose on dose on specified days
  Arms: Arm B

SUMMARY:
The purpose of this study is to assess the pharmacodynamics of Prednisolone in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations
* Body Mass Index (BMI) of 18 to 30 kilogram / square meter (kg/m2), inclusive
* Signed informed consent

Exclusion Criteria:

* Women
* Any significant acute or chronic medical illness
* Current or recent (within 3 months) gastrointestinal disease including peptic ulcer

Other protocol inclusion/exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-03-31 (Actual); Primary Completion 2008-05-05 (Actual); Study Completion 2008-05-05 (Actual)

PRIMARY OUTCOMES:
Interleukin 1 beta | Up to 32 days
  As measured by flow cytometry
Tumor necrosis factor-alpha | Up to 32 days
  As measured by flow cytometry
Receptor activator of nuclear factor-kB (RANK) | Up to 32 days
  As measured by flow cytometry
Receptor activator of nuclear factor-kB ligand (RANKL) | Up to 32 days
  As measured by flow cytometry
Osteoprotegrin (OPG) | Up to 32 days
  As measured by flow cytometry
Lipopolysaccharide Induced Cytokine Production | Up to 32 days
  As measured by blood concentration
Cell Populations | Up to 32 days
  As measured by flow cytometry
Oral glucose tolerance test | Up to 32 days
  Assessed by central labortatory
Cortisol | Up to 32 days
  As measured by the level of the hormone cortisol in the blood
Adrenocorticotropic hormone | Up to 32 days
  As measured by the level of the hormone in the blood
Osteocalcin | Up to 32 days
  As measured by blood concentration
N-terminal Pro-Collagen Peptide (PINP) | Up to 32 days
  As measured by blood concentration
Propetide type I C-term Pro-collagen Peptide (CICP) | Up to 32 days
  As measured by blood concentration
Bone-specific alkaline phosphatase | Up to 32 days
  As measured by blood concentration
Urinary deoxypyridinoline | Up to 32 days
  As measured by urine concentration
C Telopeptide of Collagen Type II (CTX-II) | Up to 32 days
  As measured by urine concentration
Calcium | Up to 32 days
  As measured by urine concentration
Creatinine | Up to 32 days
  As measured by urine concentration

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- United States (2):
  - Ppd Development, Austin, Texas
  - Local Institution, Austin, Texas

REFERENCES:
- [Derived] Hu Y, Carman JA, Holloway D, Kansal S, Fan L, Goldstine C, Lee D, Somerville JE, Latek R, Townsend R, Johnsen A, Connolly S, Bandyopadhyay S, Shadick N, Weinblatt ME, Furie R, Nadler SG. Development of a Molecular Signature to Monitor Pharmacodynamic Responses Mediated by In Vivo Administration of Glucocorticoids. Arthritis Rheumatol. 2018 Aug;70(8):1331-1342. doi: 10.1002/art.40476. Epub 2018 Jul 12. PMID 29534336